CLINICAL TRIAL: NCT04470128
Title: A Multi-center, Randomized, Two-stage, Phase II Clinical Study Evaluating the Efficacy and Safety of HSK21542 Injection for Analgesia in Subjects Undergoing Diagnostic or Therapeutic Colonoscopy
Brief Title: A Study Evaluating the Efficacy and Safety of HSK21542 Injection for Analgesia in Subjects Undergoing Colonoscopy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSK21542-202
Record Dates: First submitted 2020-07-07; First posted 2020-07-14 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Masking Description: Stage I is open-label,Stage II is double-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Stage I: HSK21542 0.5 μg/kg (Experimental): intravenous injection
  Interventions: Drug: Stage I: HSK21542 0.5 μg/kg
- Stage I: HSK21542 1 μg/kg (Experimental): intravenous injection
  Interventions: Drug: Stage I: HSK21542 1 μg/kg
- Stage II : HSK21542 0.5 μg/kg (Experimental): intravenous injection
  Interventions: Drug: HSK21542 0.5 μg/kg
- Stage II : HSK21542 1 μg/kg (Experimental): intravenous injection
  Interventions: Drug: HSK21542 1 μg/kg
- Stage II : HSK21542 2 μg/kg (Experimental): intravenous injection
  Interventions: Drug: HSK21542 2 μg/kg
- Stage II : placebo (Placebo Comparator): intravenous injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Stage I: HSK21542 0.5 μg/kg — intravenous injection
  Arms: Stage I: HSK21542 0.5 μg/kg
Drug: Stage I: HSK21542 1 μg/kg — intravenous injection
  Arms: Stage I: HSK21542 1 μg/kg
Drug: HSK21542 0.5 μg/kg — intravenous injection
  Arms: Stage II : HSK21542 0.5 μg/kg
Drug: HSK21542 1 μg/kg — intravenous injection
  Arms: Stage II : HSK21542 1 μg/kg
Drug: HSK21542 2 μg/kg — intravenous injection
  Arms: Stage II : HSK21542 2 μg/kg
Drug: Placebo — intravenous injection
  Arms: Stage II : placebo

SUMMARY:
This is a multi-center, randomized, two-stage, phase II clinical study .The main objective is to evaluate the safety and tolerability of HSK21542 injection for analgesia in patients undergoing colonoscopy, and, combining the pharmacodynamic (PD) and pharmacokinetic (PK) characteristics

ELIGIBILITY:
Inclusion Criteria:

1. Subjects undergoing diagnostic and/or therapeutic colonoscopy with an estimated operation duration of 15-45 min;
2. Aged ≥ 18 and ≤ 75 years old, with no restriction on gender;
3. American Society of Anesthesiologists (ASA) Class I-II;
4. BMI ≥ 18 kg/m^2 and ≤ 30 kg/m^2;
5. During screening and at baseline: respiratory rate ≥ 10 and ≤ 24 bpm; SpO2 ≥ 95% during inhalation; SBP ≥ 90 mmHg; DBP ≥ 50 mmHg; HR ≥ 50 and ≤ 100 bpm;
6. Subjects with intelligence and consciousness sufficient enough for cooperating with the study;
7. Capable of understanding the procedure and method of this study, willing to sign an informed consent form and to complete this study in strict accordance with the study protocol.

Exclusion Criteria:

1. Patients having contraindications to deep sedation/general anesthesia or a history of past sedation/anesthesia accidents;
2. Patients with past history of allergy or contraindications to opioids, their rescue medications, and propofol;
3. Medical history or evidence of any of the following prior to screening/at baseline, which may increase sedation/anesthesia risk:

   1. History of cardiovascular diseases: uncontrolled hypertension (systolic blood pressure [SBP] ≥ 170 mmHg and/or diastolic blood pressure [DBP] ≥ 105 mmHg without treatment, or SBP > 160 mmHg and/or DBP > 100 mmHg after antihypertensive treatment), severe arrhythmia, heart failure, Adams-Stokes syndrome, New York Heart Association (NYHA) Class ≥ III, severe superior vena cava syndrome, pericardial effusion, acute myocardial ischemia, unstable angina, myocardial infarction within 6 months before screening, history of tachycardia/bradycardia requiring medical treatment, II-III degree atrioventricular block (excluding patients with pacemakers);
   2. History of respiratory system disorders: respiratory insufficiency, history of obstructive pulmonary disease, history of bronchospasm requiring treatment within 3 months prior to screening, acute respiratory tract infection with obvious symptoms such as fever, wheezing, nasal obstruction, and cough within 1 week prior to baseline;
   3. History of neurological and psychiatric disorders: craniocerebral injury, possible convulsions, myoclonus, intracranial hypertension, cerebral aneurysms, history of cerebrovascular accidents; schizophrenia, mania, insanity, long-term use of psychotropic drugs, and history of cognitive dysfunction; history of depression, anxiety, and epilepsy, etc.;
   4. History of gastrointestinal disorders: gastrointestinal retention, active hemorrhage, or conditions that may lead to reflux and aspiration;
   5. History of alcohol abuse within 3 months prior to screening, with abuse defined as average of > 2 units of alcohol per day (1 unit = 360 mL beer or 45 mL liquor with 40% alcohol or 150 mL wine);
   6. History of drug abuse within 3 months prior to screening;
   7. History of blood donation or blood loss of ≥ 400 mL within 3 months prior to screening;
4. Patients with the following airway management risks:

   1. Asthma history, and stridor;
   2. Sleep apnea syndrome;
   3. History or family history of malignant hyperthermia;
   4. History of failed tracheal intubation;
   5. Judged by the investigator to have difficult airway or judged as difficult tracheal intubation (modified Mallampati class IV) at screening;
5. In receipt of any one of the following medications or treatments at screening:

   1. A time between the last use of opioid and non-opioid (such as paracetamol, aspirin [daily dose > 100 mg], indomethacin, diclofenac, parecoxib sodium, and other non-steroidal anti-inflammatory drugs) analgesics and randomization of shorter than 5 half-lives of the drug or the duration of the drug's efficacy (whichever is longer);
   2. Longer than 10 days of continuous use of opioid analgesics for any reason within 3 months prior to screening;
   3. Use of drugs that affect the analgesic effect within 14 days before randomization, including but not limited to: sedative-hypnotics (benzodiazepines [triazolam, diazepam, and midazolam] and non-benzodiazepines [zolpidem, zopiclone, zaleplon]), sedative-anesthetics (sevoflurane, nitrous oxide, ketamine, and etomidate), glucocorticoids (dexamethasone hydrochloride and methylprednisolone), antiepileptics (carbamazepine and sodium valproate), anxiolytics (chlordiazepoxide), antidepressants (imipramine and amitriptyline), and Chinese herbal medicines or Chinese patent medicines with analgesic and sedative effects;
   4. A time between randomization and the last use of diuretics and compound drugs containing diuretics of shorter than 5 half-lives of the drug or the duration of the drug's efficacy (whichever is longer);
6. Patient whose laboratory parameters measured at screening reach the following criteria and are verified through reexamination:

   1. WBC < 3.0 × 10^9/L;
   2. Platelet count < 80 × 10^9/L;
   3. Hemoglobin < 80 g/L;
   4. Prothrombin time > 1.5 × ULN;
   5. Activated partial thromboplastin time > 1.5 × ULN;
   6. Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≥ 2 × ULN;
   7. Total bilirubin > 1.5 × ULN;
   8. Blood creatinine > 1.5 × ULN;
7. Having participated in other drug clinical trials within 3 months prior to screening (defined as having received investigational product or placebo);
8. Pregnant or breastfeeding females: women or men of child-bearing potential who are unwilling to use contraception during the trial; subjects who are planning pregnancy within 3 months after the trial (including male subjects);
9. Subject judged by the investigator to have any other factors unsuitable for involvement in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2020-12-28 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
BPS-NI score>3 did not reach the proportion | From administration until 24 hours after administration
  the proportion of subjects with BPS-NI score>3 did not appear from the beginning of insertion of colonoscopy to the removal of colonoscopy

SECONDARY OUTCOMES:
Number of occurrences of BPS-NI score of > 3 | From administration until 24 hours after administration
  The ratio of subjects with BPS-NI scores of > 3 for 0, 1, 2, 3, or more times from the insertion to the removal of colonoscope
NRS score | From administration until 24 hours after administration
  NRS score of resting pain at each time point after the subject is fully awake
Dose of propofol used | From the first dose of the study drug to removal of colonoscope on day 1
  The total dose used during the induction period, maintenance period, and the entire study process
Success rate of colonoscopy diagnosis and treatment | From the first dose of the study drug to removal of colonoscope on day 1
  The following two conditions must be met for successful diagnosis and treatment:
  complete colonoscopy diagnosis and treatment and failure to use remedial analgesics
Time to full recovery | On day 1
  The time from the removal of colonoscope to when the subject opens his/her eyes and can tell his/her date of birth
Time to discharge | On day 1
  The time from the removal of colonoscope to the occurrence of 3 consecutive Aldrete score of ≥ 9
The incidence and severity of AEs | from signing the informed consent form to the follow-up period
  Adverse event/serious adverse event

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, China